CLINICAL TRIAL: NCT02812771
Title: A Multicenter, Open Label, Single-arm Study Evaluating the Safety and Pharmacokinetics of Efinaconazole Topical Solution in Subjects With Mild to Severe Onychomycosis of the Toenails
Brief Title: Safety and Pharmacokinetics of Efinaconazole Topical Solution in Subjects With Mild to Severe Onychomycosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-108A-401
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — efinaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Efinaconazole (Experimental): Efinaconazole
  Interventions: Drug: Efinaconazole

INTERVENTIONS:
Drug: Efinaconazole — Solution

SUMMARY:
Safety and Pharmacokinetics (PK) of a once daily topical application of efinaconazole in the treatment of pediatric subjects with mild to severe onychomycosis of the toenails.

DETAILED DESCRIPTION:
This is an open label, single-arm study designed to evaluate the safety and PK of a once daily topical application of efinaconazole in the treatment of pediatric subjects with mild to severe onychomycosis of the toenails.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects of any race, 6 to 16 years of age (inclusive). PK Subset: Male or female subjects of any race, 12 to 16 years of age (inclusive).
* Verbal and written informed consent/assent obtained from the subject and/or their parent or legal guardian.
* Good general health, as assessed by the investigator, based on the subject's medical history, physical examination, and safety laboratory tests.
* Target great toenail for all subjects, and both great toenails for subjects in the PK subset, must have evidence of toenail growth, per subject's report that monthly clipping is needed.
* Subjects and their parents/legal guardians are willing to comply with study instructions and return to the investigational center for all required visits (a visit schedule with the length of each visit will be provided to ensure that the subject can meet the requirements and have adequate transportation).

Key Exclusion Criteria:

* Females who are pregnant, nursing an infant, or planning a pregnancy during the study period.
* History of immunosuppression and/or clinical signs indicative of possible immunosuppression, as determined by the investigator, or known human immunodeficiency virus infection.
* History of diabetes that is uncontrolled as determined by the investigator (diabetes that is controlled by diet or medication does not exclude a subject).
* Presence of any toenail infection other than or in addition to dermatophytes, such as Scytalidium as determined by the investigator (candidal onychomycosis infection, concurrent with a positive dermatophyte culture, is acceptable).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu Alexander, MD, Study Director — Valeant Pharmaceuticals
Locations (10):
- United States (9):
  - Valeant Site 01, Birmingham, Alabama
  - Valeant Site 04, Fountain Valley, California
  - Valeant Site 03, Santa Rosa, California
  - Valeant SIte 05, South Miami, Florida
  - Valeant Site 09, New Orleans, Louisiana
  - Valeant Site 08, Baltimore, Maryland
  - Valeant Site 02, Forest Hills, New York
  - Valeant Site 06, Philadelphia, Pennsylvania
  - Valeant Site 07, McAllen, Texas
- Valeant Site 10, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efinaconazole
Started | 62
Completed | 50
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Of the 62 participants who were enrolled in the study, 2 did not apply study drug and were excluded from all analysis populations.
Arm/Group | Efinaconazole
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 53
  More than one race | 0
  Unknown or Not Reported | 1
Target Great Tonail [Count of Participants; unit: Participants]
  Left | 32
  Right | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Adverse Event
Time Frame: 48 weeks
Population: All participants who received at least 1 confirmed dose of study drug (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Efinaconazole
Number analyzed (Participants) | 60
Participants | 39

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: All participants who received at least 1 confirmed dose of study drug (Safety Population).
Arm/Group | Efinaconazole
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 20/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efinaconazole (N=60)
Pneumonia (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efinaconazole (N=60)
Food poisoning (Gastrointestinal disorders) | 3
Influenza (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 4
Nail injury (Injury, poisoning and procedural complications) | 4
Headache (Nervous system disorders) | 6
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4
Nasopharyngitis (Infections and infestations) | 18
Tinea pedis (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02812771/Prot_SAP_000.pdf